CLINICAL TRIAL: NCT05035225
Title: A National Survey on the Prevalence and Impact of Multiple Pharmacy Use in Specialty Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Illinois at Chicago (Other); University of California, Los Angeles (Other); University of Washington (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00277792
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Health Services Accessibility
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specialty Pharmacy Patient (Experimental): Patients who have been prescribed at least one selected specialty medication
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Multiple Pharmacy Use Survey

SUMMARY:
Specialty medications often have dispensing restrictions which can be dictated by manufacturer limited distribution strategies, narrow insurance networks, or a combination of both. Unfortunately, this may result in patients being required to use 2 or more pharmacies to fill their prescription medications; this is referred to as multiple pharmacy use (MPU). The investigators' plan is to administer a survey to patients who have been prescribed one or more specialty medications to evaluate the prevalence of MPU in this population as well as to investigate patients' attitudes about MPU and potential factors increasing the likelihood of MPU

DETAILED DESCRIPTION:
The investigators will identify patients from participating member sites via a review of prescribing records for specific specialty medications. Patients will be contacted via telephone to explain the purpose and risk of the study. Consented patients will then be asked a series of 11 questions about their attitudes and experience with taking and obtaining their specialty medication(s). Additional demographic and clinical information about patients will be collected via chart review.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* English-speakers
* An active patient of a performance institution and ability to provide informed consent to participate with the survey
* Electronically prescribed at least one specialty medication by a performance site provider, which can be either a new or renewed order, within the last 3 months

Exclusion Criteria:

* Subjects less than 18 years of age
* Non-English speakers
* Patients that cannot or are unwilling to provide consent
* Patients who have not had a new or renewed specialty medication prescription order placed electronically within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients using Multiple Pharmacies | Within one year of study initiation
  Of all patients consented, the percentage of patients using more than one pharmacy to obtain their medications

SECONDARY OUTCOMES:
Self-reported adherence and barriers | Within one year of study initiation
  Patient response to questions about having missed doses in the past month
Method of obtaining medications | Within one year of study initiation
  Patient response to questions about distance from pharmacy and how prescriptions are primarily obtained
Experience with obtaining and administering medications | Within one year of study initiation
  Patient response to questions about how easy it is for patients to obtain and administer medication

CONTACTS AND LOCATIONS:
Overall Officials: Whisler, PharmD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data from individual study sites will be collected and stored together either via a password-protected Excel file or Qualtrics.